CLINICAL TRIAL: NCT05856435
Title: Tailoring the Chicago Parent Program for the Foster Care Setting
Brief Title: Tailoring CPP for the Foster Care Setting
Acronym: CPP-FC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Johns Hopkins University (Other); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0228
Record Dates: First submitted 2023-04-17; First posted 2023-05-12 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Behavior Problem
Keywords: foster care; child behavior; parenting skills; behavioral health
MeSH Terms: conditions — Mental Disorders; Child Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chicago Parent Program for Foster Care (Other): Caregiver parent training sessions.
  Interventions: Behavioral: Chicago Parent Program for Foster Care

INTERVENTIONS:
Behavioral: Chicago Parent Program for Foster Care — The Chicago Parent Program for Foster Care FC consists of a 12-session parent training program that focuses on building caregiver-child relationships, behavioral management strategies, managing caregiver stress, and skill maintenance.

SUMMARY:
The primary objective of this study is to tailor the Chicago Parent Program, an evidence-based parent training program, for the foster care setting and pilot the content in two cohorts of foster and kinship caregivers (Gross et al., 2009).

DETAILED DESCRIPTION:
This study involves the administration of an evidence-based prevention program to prevent and reduce behavior problems in young children (the Chicago Parent Program; CPP). CPP will be tailored by creating additional handouts, discussion questions, and topics that contextualize CPP material to foster care, to meet the needs and social norms of foster and kinship caregivers. The CPP-FC 12-session curriculum will be delivered to two cohorts of foster and kinship caregivers virtually. Data for this study will come from multiple sources, including caregiver participant report and a review of existing electronic databases at CCHMC.

ELIGIBILITY:
Inclusion Criteria:

* Must be a licensed foster caregiver or kinship caregiver to a child ages 2 years to 8 years
* Must be in good standing with the foster care agency
* Must be English-speaking

Exclusion Criteria:

* Not having a foster child ages 2 - 8 years in the home
* Caregiver is unable to commit to participating in CPP-FC
* This foster child age 2 - 8 years was placed in the home more than 45 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2027-08-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Beal, PhD, Principal Investigator — Cincinnati Children's Hospital Medical Center Cincinnati, OH USA
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee EH. Review of the psychometric evidence of the perceived stress scale. Asian Nurs Res (Korean Soc Nurs Sci). 2012 Dec;6(4):121-7. doi: 10.1016/j.anr.2012.08.004. Epub 2012 Sep 18. PMID 25031113
- [Background] Guo M, Morawska A, Filus A. Initial Validation of the Parent-Report Child Adjustment and Parent Efficacy Scale (CAPES) in a Chinese Cultural Context. Assessment. 2018 Dec;25(8):1056-1073. doi: 10.1177/1073191116681493. Epub 2016 Dec 20. PMID 30392414
- [Background] Heerman WJ, Taylor JL, Wallston KA, Barkin SL. Parenting Self-Efficacy, Parent Depression, and Healthy Childhood Behaviors in a Low-Income Minority Population: A Cross-Sectional Analysis. Matern Child Health J. 2017 May;21(5):1156-1165. doi: 10.1007/s10995-016-2214-7. PMID 28092060
- [Background] Gross D, Fogg L, Young M, Ridge A, Cowell J, Sivan A, Richardson R. Reliability and validity of the Eyberg Child Behavior Inventory with African-American and Latino parents of young children. Res Nurs Health. 2007 Apr;30(2):213-23. doi: 10.1002/nur.20181. PMID 17380522
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] Agazio JB, Buckley KM. Revision of a Parental Stress Scale for use on a pediatric general care unit. Pediatr Nurs. 2012 Mar-Apr;38(2):82-7. PMID 22685867
- [Background] Wilson PA, Hansen NB, Tarakeshwar N, Neufeld S, Kochman A, Sikkema KJ. SCALE DEVELOPMENT OF A MEASURE TO ASSESS COMMUNITY-BASED AND CLINICAL INTERVENTION GROUP ENVIRONMENTS. J Community Psychol. 2008 Apr;36(3):271-288. doi: 10.1002/jcop.20193. PMID 19018295
- [Background] Gross D, Garvey C, Julion W, Fogg L, Tucker S, Mokros H. Efficacy of the Chicago parent program with low-income African American and Latino parents of young children. Prev Sci. 2009 Mar;10(1):54-65. doi: 10.1007/s11121-008-0116-7. PMID 19067166

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on the age of an index foster child and the duration of placement of the foster child at two foster care consultation clinic locations within a single academic medical center between May 2023 and July 2023. The first participant was enrolled on May 16, 2023, and the last participant was enrolled on July 14, 2023.
Period: Overall Study
Arm/Group | Chicago Parent Program for Foster Care
Started | 16
Completed | 10
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Chicago Parent Program for Foster Care
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.43 (15.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 6
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 16
Perceived Stress Scale [Mean (Standard Deviation); unit: units on a scale] — The Perceived Stress Scale is a 14-item self-report measure of how unpredictable, uncontrollable, and overloaded individuals find their life circumstances. All items are rated on a 5-point scale, ranging from 0 ("Never") to 4 ("very often"). Some items are reverse-scored. Responses are summed to yield a total score (range 0 - 56), with higher scores indicating greater perceived stress.
  units on a scale | 16.44 (8.30)
Child Adjustment & Parent Efficacy Scale [Mean (Standard Deviation); unit: units on a scale] — The Child Adjustment & Parent Efficacy Scale, Total Intensity subscale is a 27-item measure of child behavior and emotional problems. Item responses are rated on a 4-point scale, ranging from 0 ("Not true of my child at all") to 3 ("True of my child very much"/"Most of the time"). Twenty-four items are summed to yield a Behavior Problems score (range 0-72), and three items are summed to yield an Emotional Problems score (range 0-9). Behavioral and Emotional Problems scores can be summed for a Total Intensity score (range 0-81). Higher scores indicate a higher level of problems.
  units on a scale
    Behavior Problems Scale | 25.74 (17.12)
    Emotional Problems Scale | 2.06 (1.37)
    Total Intensity Scale | 27.79 (18.63)
Parenting Sense of Competence Scale [Mean (Standard Deviation); unit: units on a scale] — The Parenting Sense of Competence Scale is a 17-item questionnaire that measures overall parenting satisfaction and competence. Items are measured on a 6-point scale, with responses ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"). Some items are reverse-scored. Items are summed to yield a total scale (range 17-102) and two subscales: parental self-efficacy (range 8-48) and parental satisfaction (range 9-54). Higher scores indicate higher levels of parental self-efficacy and parental satisfaction.
  units on a scale
    Parental Satisfaction Scale | 38.33 (7.99)
    Parental Self-Efficacy Scale | 35.25 (6.31)
    Total Scale | 73.98 (12.09)
Eyberg Child Behavior Inventory [Mean (Standard Deviation); unit: T-score] — The Eyberg Child Behavior Inventory, a 36-item measure that assesses child behavior problems. Each item has 2 parts that make up 2 subscales: Intensity and Problem. Intensity items are rated on a 7-point scale, from 1 (Never) to 7 (Always), and Problem items are Yes/No responses. Items from each scale are summed to yield raw scores and converted to T-scores (M=50, SD=10). Higher Intensity scores indicate more frequent displays of the child behaviors, and higher Problem scores indicate the parent perceives the behaviors as more problematic. T-scores above 60 indicate elevated behavior problems.
  T-score
    Intensity Scale T-Score | 53.00 (13.73)
    Problem Scale T-Score | 47.19 (10.04)
Parental Stress Scale [Mean (Standard Deviation); unit: units on a scale] — The Parental Stress Scale is an 18-item questionnaire that assesses parental stress relating to parental sensitivity to the child, child behavior, and quality of the parent-child relationship. Items are rated on a 5-point scale, ranging from 1 ("Strongly disagree") to 5 ("Strongly agree"). Some items are reverse-scored. Items are summed to yield a total score (range 18-90), with higher scores indicating higher levels of parental stress.
  units on a scale | 34.56 (11.90)

OUTCOME MEASURES:

1. Primary Outcome: Change in Perceived Stress Scale
Description: The Perceived Stress Scale is a 14-item self-report measure of how unpredictable, uncontrollable, and overloaded individuals find their life circumstances. All items are rated on a 5-point scale, ranging from 0 ("Never") to 4 ("very often"). Some items are reverse-scored. Responses are summed to yield a total score (range 0 - 56), with higher scores indicating greater perceived stress.
Time Frame: Pre Intervention and 18 weeks
Population: N = 16 participants completed the Perceived Stress Scale at Pre Intervention and n = 10 participants completed the Perceived Stress Scale at 18 Weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chicago Parent Program for Foster Care
Number analyzed (Participants) | 16
score on a scale
  Sample Mean at 18 Weeks: number analyzed (Participants) | 10
  Sample Mean at 18 Weeks | 14.70 (8.41)
  Mean Difference from Pre Intervention to 18 Weeks | 0.20 (8.78)

2. Primary Outcome: Change in Child Adjustment & Parent Efficacy Scale
Description: The Child Adjustment & Parent Efficacy Scale, Total Intensity subscale is a 27-item measure of child behavior and emotional problems. Item responses are rated on a 4-point scale, ranging from 0 ("Not true of my child at all") to 3 ("True of my child very much"/"Most of the time"). Twenty-four items are summed to yield a Behavior Problems score (range 0-72), and three items are summed to yield an Emotional Problems score (range 0-9). Behavioral and Emotional Problems scores can be summed for a Total Intensity score (range 0-81). Higher scores indicate a higher level of problems.
Time Frame: Pre Intervention and 18 weeks
Population: N = 16 participants completed The Child Adjustment & Parent Efficacy Scale at Pre Intervention and n = 10 participants completed The Child Adjustment & Parent Efficacy Scale at 18 Weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chicago Parent Program for Foster Care
Number analyzed (Participants) | 16
score on a scale
  Total Intensity Scale Sample Mean at 18 Weeks: number analyzed (Participants) | 10
  Total Intensity Scale Sample Mean at 18 Weeks | 24.61 (15.63)
  Total Intensity Scale Mean Difference from Pre Intervention to 18 Weeks | -4.59 (14.83)
  Behavior Problems Scale Sample Mean at 18 Weeks: number analyzed (Participants) | 10
  Behavior Problems Scale Sample Mean at 18 Weeks | 24.52 (14.80)
  Behavior Problems Scale Mean Difference from Pre Intervention to 18 Weeks | -4.18 (14.27)
  Emotional Problems Scale Sample Mean at 18 Weeks: number analyzed (Participants) | 10
  Emotional Problems Scale Sample Mean at 18 Weeks | 1.90 (1.37)
  Emotional Problems Scale Mean Difference from Pre Intervention to 18 Weeks | -0.40 (1.17)

3. Primary Outcome: Change in Parenting Sense of Competence Scale
Description: The Parenting Sense of Competence Scale is a 17-item questionnaire that measures overall parenting satisfaction and competence. Items are measured on a 6-point scale, with responses ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"). Some items are reverse-scored. Items are summed to yield a total scale (range 17-102) and two subscales: parental self-efficacy (range 8-48) and parental satisfaction (range 9-54). Higher scores indicate higher levels of parental self-efficacy and parental satisfaction.
Time Frame: Pre Intervention and 18 weeks
Population: N = 16 participants completed the Parenting Sense of Competence Scale at Pre Intervention and n = 10 participants completed the Parenting Sense of Competence Scale at 18 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chicago Parent Program for Foster Care
Number analyzed (Participants) | 16
score on a scale
  Total Scale Sample Mean at 18 Weeks: number analyzed (Participants) | 10
  Total Scale Sample Mean at 18 Weeks | 72.60 (10.70)
  Total Scale Mean Difference from Pre Intervention to 18 Weeks | -0.10 (11.63)
  Parental Satisfaction Scale Sample Mean at 18 Weeks: number analyzed (Participants) | 10
  Parental Satisfaction Scale Sample Mean at 18 Weeks | 38.50 (8.42)
  Parental Satisfaction Mean Difference from Pre Intervention to 18 Weeks | 0.70 (6.38)
  Parental Self-Efficacy Scale Sample Mean at 18 Weeks: number analyzed (Participants) | 10
  Parental Self-Efficacy Scale Sample Mean at 18 Weeks | 34.10 (7.67)
  Parental Self-Efficacy Mean Difference from Pre Intervention to 18 Weeks | -0.80 (8.68)

4. Primary Outcome: Change in Eyberg Child Behavior Inventory
Description: The Eyberg Child Behavior Inventory, a 36-item measure that assesses child behavior problems. Each item has 2 parts that make up 2 subscales: Intensity and Problem. Intensity items are rated on a 7-point scale, from 1 (Never) to 7 (Always), and Problem items are Yes/No responses. Items from each scale are summed to yield raw scores and converted to T-scores (M=50, SD=10). Higher Intensity scores indicate more frequent displays of the child behaviors, and higher Problem scores indicate the parent perceives the behaviors as more problematic. T-scores above 60 indicate elevated behavior problems.
Time Frame: Pre Intervention and 18 weeks
Population: N = 16 participants completed The Eyberg Child Behavior Inventory at Pre Intervention and n = 10 participants completed The Eyberg Child Behavior Inventory at 18 Weeks.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Chicago Parent Program for Foster Care
Number analyzed (Participants) | 16
T-score
  Intensity Scale T-Score Sample Mean at 18 Weeks: number analyzed (Participants) | 10
  Intensity Scale T-Score Sample Mean at 18 Weeks | 53.70 (12.49)
  Intensity Scale T-Score Mean Difference from Pre Intervention to 18 Weeks | -2.10 (10.24)
  Problem Scale T-Score Sample Mean at 18 Weeks: number analyzed (Participants) | 10
  Problem Scale T-Score Sample Mean at 18 Weeks | 48.80 (6.97)
  Problem Scale T-Score Mean Difference from Pre Intervention to 18 Weeks | 0.50 (9.63)

5. Primary Outcome: Strengths and Difficulties Questionnaire
Description: The Strengths and Difficulties Questionnaire (SDQ) is a 25-item questionnaire that assesses child behavior. Items are rated on a 3-point scale and responses range from 0 ("Not true") to 2 ("Certainly true"). Some items are reverse-scored. Items are summed to yield 5 subscales: Emotional Problems, Conduct Problems, Hyperactivity, Peer Problems, and Prosocial (ranges 0 -10). A total score (range 0-40) is calculated using the sum of all the subscales, except Prosocial. Higher scores in each subscale and the total score indicate more child behavior problems.
Time Frame: Pre Intervention and 18 weeks
Population: N = 10 participants completed The Strengths and Difficulties Questionnaire at 18 Weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chicago Parent Program for Foster Care
Number analyzed (Participants) | 10
score on a scale
  Emotional Problems Scale Sample Mean at 18 Weeks | 2.40 (2.22)
  Conduct Problems Scale Sample Mean at 18 Weeks | 2.60 (1.96)
  Hyperactivity Scale Sample Mean at 18 Weeks | 5.70 (3.47)
  Peer Problems Scale Sample Mean at 18 Weeks | 3.60 (1.84)
  Prosocial Problems Scale Sample Mean at 18 Weeks | 6.00 (2.05)
  Total Scale Sample Mean at 18 Weeks | 14.30 (7.76)

6. Primary Outcome: Change in Parental Stress Scale
Description: The Parental Stress Scale is an 18-item questionnaire that assesses parental stress relating to parental sensitivity to the child, child behavior, and quality of the parent-child relationship. Items are rated on a 5-point scale, ranging from 1 ("Strongly disagree") to 5 ("Strongly agree"). Some items are reverse-scored. Items are summed to yield a total score (range 18-90), with higher scores indicating higher levels of parental stress.
Time Frame: Pre Intervention and 18 weeks
Population: N = 16 participants completed The Parental Stress Scale at Pre Intervention and n = 10 participants completed The Parental Stress Scale at 18 Weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chicago Parent Program for Foster Care
Number analyzed (Participants) | 16
score on a scale
  Total Scale Sample Mean at 18 Weeks: number analyzed (Participants) | 10
  Total Scale Sample Mean at 18 Weeks | 36.00 (12.24)
  Total Scale Mean Difference from Pre Intervention to 18 Weeks | 0.80 (4.47)

7. Primary Outcome: Change in Group Environment Scale
Description: The Group Environment Scale is a 25-item measure that assesses the dimensions of intervention group environments. Items are rated on a 5-point scale, with responses ranging from 1 ("Strongly disagree") to 5 ("Strongly agree"). Items are averaged to yield three subscales: Cohesiveness, Implementation and Preparedness, and Counterproductive Activity. Higher scores on the Cohesiveness Scale (range 1-5) indicate more group cohesiveness. Higher scores on the Implementation and Preparedness Scale (range 1-5) indicate greater group implementation quality. Higher scores on the Counterproductive Activity Scale (range 1-5) indicate more counterproductive group activities.
Time Frame: Week 7, Week 11, Week 19
Population: N = 2 participants completed The Group Environment Scale at Week 7, n = 4 participants completed The Group Environment Scale at Week 11, and n = 7 participants completed The Group Environment Scale at Week 19.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chicago Parent Program for Foster Care
Number analyzed (Participants) | 7
score on a scale
  Cohesiveness Scale Sample Mean at 7 Weeks: number analyzed (Participants) | 2
  Cohesiveness Scale Sample Mean at 7 Weeks | 4.44 (0.44)
  Cohesiveness Scale Sample Mean at 11 Weeks: number analyzed (Participants) | 4
  Cohesiveness Scale Sample Mean at 11 Weeks | 4.48 (0.40)
  Cohesiveness Scale Sample Mean at 19 Weeks | 4.30 (0.51)
  Cohesiveness Scale Mean Difference from 7 Weeks to 11 Weeks: number analyzed (Participants) | 4
  Cohesiveness Scale Mean Difference from 7 Weeks to 11 Weeks | 0.19 (0.09)
  Cohesiveness Scale Mean Difference from 11 Weeks to 19 Weeks | 0.16 (0.52)
  Implementation and Preparedness Scale Sample Mean at 7 Weeks: number analyzed (Participants) | 2
  Implementation and Preparedness Scale Sample Mean at 7 Weeks | 4.55 (0.26)
  Implementation and Preparedness Scale Sample Mean at 11 Weeks: number analyzed (Participants) | 4
  Implementation and Preparedness Scale Sample Mean at 11 Weeks | 4.71 (0.55)
  Implementation and Preparedness Scale Sample Mean at 19 Weeks | 4.40 (0.52)
  Implementation and Preparedness Scale Mean Difference from 7 Weeks to 11 Weeks: number analyzed (Participants) | 4
  Implementation and Preparedness Scale Mean Difference from 7 Weeks to 11 Weeks | 0.41 (0.19)
  Implementation and Preparedness Scale Mean Difference from 11 Weeks to 19 Weeks | 0.11 (0.75)
  Counterproductive Activity Scale Sample Mean at 7 Weeks: number analyzed (Participants) | 2
  Counterproductive Activity Scale Sample Mean at 7 Weeks | 4.83 (0.24)
  Counterproductive Activity Scale Sample Mean at 11 Weeks: number analyzed (Participants) | 4
  Counterproductive Activity Scale Sample Mean at 11 Weeks | 4.77 (0.32)
  Counterproductive Activity Scale Sample Mean at 19 Weeks | 4.43 (0.79)
  Counterproductive Activity Scale Mean Difference from 7 Weeks to 11 Weeks: number analyzed (Participants) | 4
  Counterproductive Activity Scale Mean Difference from 7 Weeks to 11 Weeks | -0.42 (0.35)
  Counterproductive Activity Scale Mean Difference from 11 Weeks to 19 Weeks | 0.04 (0.48)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for approximately 19 weeks that each participant was enrolled.
Description: Adverse event data were collected in a non-sytematic approach for enrolled participants. This is a minimal-risk study which involves an evidence-based behavioral intervention, and no adverse events were expected to occur.
Arm/Group | Chicago Parent Program for Foster Care
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
Due to an error in survey firing logic, The Strength and Difficulties Questionnaire was not administered at the Pre Intervention event. There are only sample means for the scale scores, and no mean differences listed in Outcome Measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT05856435/Prot_SAP_002.pdf
  • Informed Consent Form (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT05856435/ICF_001.pdf